CLINICAL TRIAL: NCT02810054
Title: Periodontal Minimally Invasive Surgical Techniques With or Without Enamel Matrix Derivative Gel for Treatment of Intrabony Periodontal Osseous Defects in Humans.
Brief Title: Using MIST With or Without EMD in Treatment of Intrabony Periodontal Defects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Muataz Osman, Dr, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSCPERIO-001
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Intrabony Periodontal Defects
Keywords: regeneration; intrabony defects; enamel matrix derivative; MIST

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (MIST without EMD) (Sham Comparator): Those participants who will receive the minimally invasive surgical techniques but without application Enamel Matrix Derivative (EMD) .
  Interventions: Procedure: Minimally Invasive Surgical Techniques (MIST)
- Test Group (MIST with EMD) (Experimental): Those participant who will receive the minimally invasive surgical techniques with the application of Enamel Matrix Derivative (EMD) .
  Interventions: Procedure: Minimally Invasive Surgical Techniques (MIST); Procedure: Enamel Matrix Derivative (EMD)

INTERVENTIONS:
Procedure: Minimally Invasive Surgical Techniques (MIST) — Using minimally invasive surgical techniques.
Procedure: Enamel Matrix Derivative (EMD) — Use of enamel matrix derivative for the treatment of intrabony periodontal defects.
  Arms: Test Group (MIST with EMD)

SUMMARY:
After performing the power calculation, healthy adult participants for the study will be randomly allocated into two groups. The intervention group will receive minimally invasive surgical techniques (MIST) with enamel matrix derivative (Emdogain) as a treatment of intrabony periodontal defect. The control group will receive minimally invasive surgical techniques (MIST) without enamel matrix derivative (Emdogain).

Clinical attachment level (CAL) gain and periodontal pocket depth (PPD) reduction as well as the position of gingival margin (REC) as the main outcomes and the radiographic intrabony infill, bleeding on probing (BoP), full mouth plaque score (FMPS) and full mouth bleeding score (FMBS) as secondary outcome will be recorded for the participants by 3 examiners at three stages:

1. Before the procedure as a baseline record.
2. 6 months after surgery, all parameters EXCEPT intra oral periapical (PA) radiographs.
3. 12 months after surgery.

The readings will be recorded using The University of Michigan O Probe with William's Calibration OR Pressure Sensitive Periodontal Probe at 0.3 N to the nearest millimeter for the clinical attachment level gain (CAL), the periodontal pocket depth (PPD) and the position of gingival margin (REC), present or absent for the bleeding on probing (BoP), and intra oral periapical (PA) radiograph for crestal bone level assessment.

DETAILED DESCRIPTION:
The surgical procedure appointment will take probably 45-75 minutes. The procedures will take the following steps:

1. One Intra-oral periapical radiograph/X-ray should have been taken before the procedure and another one at month 12.
2. Providing local anesthetics to numb the area to be worked on and it is just for selected sites and no need for general anesthesia at all.
3. Using micro surgical blade to cut the gum very conservatively, as we will be using a very conservative minimally invasive surgical technique up-to-date.
4. After establishing the visibility to the defective site with help of dental loups as a part of the procedure, we will clean the whole area using manual and ultrasonic cleaning instrument and making sure that there is no granulation (infected/inflamed) tissue inside the defect and the root surfaces of the affected tooth/teeth are very smooth.
5. In case of using enamel matrix derivative gel (Emdogain) we will apply the material as the manufacturer recommends, while in the case of not using the enamel matrix derivative gel (Emdogain) we will do the standard open flap debridement (OFD) scaling and root planning for the affected sites and then closing and securing the flap/wound with exactly the same minimally invasive surgical technique.
6. According to the technique to be used we will use the suitable type of suture material and technique to make sure that the flap/wound is closed in place and secured properly.
7. At the end of the procedure the patient will receive post-operative instructions which are a kind of Do's & Don't as follow:

   A. Don't clean the wound for the next 2 weeks. B. Using chlorhexidine based mouth wash 0.12% twice a day for 3 weeks. C. Don't eat or drink hot food and drinks for the first 2 days, after that you may start using warm food and back to normal in a week time.

   C. Don't play or disturb the suture with your tongue, lips or fingers. D. Try not to do exercises during the 1st week. E. Do brush the rest of your teeth.
8. The participant will be asked to attend a 15 minutes appointment 7-10 days right after the procedure for suture removal. Then every two weeks until month 3 just for evaluation of healing and performing any kind of treatment that might be needed for example; superficial cleaning. Then you will be asked to attend one appointment a month until month 6 to take the measurements again and providing any cleaning needed, then at month 9, and finally, at month 12 to take the measurements for the last time to compare them with the baseline measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate from both gender males and females with moderate to advanced periodontal disease.
2. 18 years old and more.
3. Probing pocket depth (PPD) of > 5mm and clinical attachment loss (CAL) of >6mm.
4. 2 and 3-wall angular intra bony periodontal defects.
5. Full-mouth plaque score (FMPS) of < 20%.
6. Full-mouth bleeding score (FMBS) of < 15%.
7. Medically fit and healthy.
8. Not allergic to any materials or medications that could be used during or after the procedure.

Exclusion Criteria:

1. Patients with diabetes and any haematological disorders that might compromise the procedure.
2. 1-wall and crater defects.
3. Immunocompromised patients and those with known allergy to one of the materials or medications to be used.
4. Patients whose FMPS > 20%.
5. Smokers.
6. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
clinical attachment level gain CAL | 12 months
  periodontal clinical attachment level gain

SECONDARY OUTCOMES:
radiographic bone fill | 12 months
  assessing the bone level from the cemento-enamel junction to the crestal bone height
full mouth bleeding score FMBS | 12 months
full mouth dental plaque score FMPS | 12 months
periodontal probing depth reduction PPD | 12 months
marginal gingival recession REC | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Seymour, Study Director — The University of Manchester

IPD SHARING:
Plan to Share IPD: No
Individual Participant data will not be shared however once anonymised the results may be published.